CLINICAL TRIAL: NCT02705950
Title: Effect of Intrathecal Baclofen (ITB) Bolus on Neuropathic Pain (NP) in Spinal Cord Injury (SCI) Patients. Preliminary Study.
Brief Title: Intrathecal Baclofen (ITB) Bolus on Neuropathic Pain (NP). Preliminary Study.
Acronym: ITB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Guttmann (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Hatice Kumru, MD PhD, Institut Guttmann
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014187
Record Dates: First submitted 2016-02-25; First posted 2016-03-11 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intrathecal baclofen bolus (Active Comparator): In ITB bolus group: An intrathecal baclofen bolus injection of 50 µg (1ml) will be injected at L3/L4 level. A 50 µg.
  Interventions: Drug: Intrathecal baclofen bolus
- placebo (Placebo Comparator): In the placebo group: 1 ml of physiological saline (isotonic saline) will be injected subcutaneously at L3/L4 level simulating
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Intrathecal baclofen bolus — An intrathecal baclofen bolus injection of 50 µg (1ml) will be injected at L3/L4 level.
  Other Names: ITB bolus
  Arms: intrathecal baclofen bolus
Other: Placebo — 1 ml of physiological saline (isotonic saline) will be injected subcutaneously at L3/L4 level simulating
  Other Names: physiological saline
  Arms: placebo

SUMMARY:
Hypothesis:

ITB bolus can have antinociceptive effect on neuropathic pain in spinal cord injury patients, which could depend on the subtype of pain, or on the lesion level, cervical or thoracic spinal cord injury.

Objective:

To study the effect of intrathecal baclofen bolus on neuropathic pain in patients with spinal cord injury at cervico-dorsal level.

Primary Endpoint:

Effect of intrathecal baclofen bolus in neuropathic pain (measured using the Neuropathic Pain Inventory Scale, the Brief Pain Inventory and the Numerical Rating Scale) in spinal cord injury at cervico-dorsal level.

Secondary Endpoints:

1. Spasticity and spasms (measured using the Modified Ashworth Scale and the Visual Analogue Scale and Penn Spasm Frequency Scale).
2. Neurophysiological examination (warm perception threshold, heat pain perception threshold, evoked pain perception and contact heat evoked potentials).

DETAILED DESCRIPTION:
The study will be a randomized, double-blind (patients and who will realize the clinical and neurophysiologic evaluation), placebo-controlled trial. We will recruit 10-12 patients with SCI with complete or incomplete lesion at cervical or thoracic level to be randomly distributed in two study groups: ITB bolus group and a placebo group.

In 6-8 months, we will administer an intrathecal baclofen bolus of 50 µg (1ml) in 5-6 SCI patients or 1ml of physiologic serum subcutaneously in the other 5-6 SCI patients.

Before the intrathecal baclofen or placebo bolus is administered, patients will be evaluated for neuropathic pain, using the Neuropathic Pain Inventory Scale, Brief Pain Inventory and Numerical Rating Scale. Spasticity and spasms will also be measured by the Modified Ashworth Scale, the Visual Analogue Scale and the Penn Spasm. After that, patients will also undergo, early in the morning when the intrathecal baclofen or placebo bolus will be administered, a neurophysiology assessment (warm perception threshold, heat pain perception threshold, evoked pain perception and contact heat evoked potentials).

After the neurophysiological evaluation, patients will receive an intrathecal baclofen bolus of 50 µg or placebo (randomization). After the intrathecal baclofen or placebo injection, a clinical and neurophysiological examination, of neuropathic pain and spasticity and spasms, will be repeated at 1, 2 and 4 hours after the bolus administration. Moreover, Kumru et al. (2013) reported that the 50 µg intrathecal baclofen bolus reduced the pain perception threshold and evoked acute pain perception in patients with SCI.

During all evaluation period, the patients continue with their analgesic, antispastic and/or any other stable medication.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years and at least one year since the spinal cord injury.
* Aetiology: stable SCI from traumatic or medical origin.
* Patients with chronic refractory neuropathic pain and with spinal cord injury, both complete and incomplete, at the cervico-thoracic level.
* Severity of pain equal or greater than 4 in the Numerical Rating Scale.
* With spasticity (MAS>=).
* Stable analgesic, antispastic and any other medication.

Exclusion Criteria:

* Patients who do not give patient inform consent.
* Contraindication for baclofen or intrathecal injection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Neuropathic Pain Inventory Scale (NPIS) | Change from baseline in neuropathic pain at 4hours
  a self-questionnaire specifically designed to evaluate the different symptoms of neuropathic pain and includes 10 descriptors that allow discrimination and quantification of five distinct clinically relevant dimensions of neuropathic pain syndromes and that are sensitive to treatment

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | Change from baseline in spasticity at 1, 2 and 4hours
  is to measure spasticity in patients who have lesions of the central nervous system or neurological disorders.
Modified Penn Spasm Frequency Scale | Change from baseline in spasticity at 4hours
  2 component self-report measure of the frequency of reported muscle spasms which is commonly used to quantify spasticity.
Visual Analogue Scale (VAS) for spasticity | Change from baseline in spasticity at 4 hours
  Consists 10cm line for patient self-reporting of spasticity last 24hours
warm and heat pain perception threshold | Change from baseline in warm and pain perception at 4hours
  it is quantitative sensory perception test for warm perception threshold and heat pain perception threshold
evoked pain perception | Change from baseline in evoked acute pain perception at 4hours
  it is quantitative sensory perception test for acute induced pain perception measurement
contact heat evoked potentials. | Change from baseline in evoked potential with heat pain at 4hours
  It is an evoked potential induced with heat painful stimulus
Brief Pain Inventory (BPI) | Change from baseline in pain at 4hours
  The BPI allows patients to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function.
Numerical Rating Scale (NRS) for neuropathic pain | Change from baseline in pain at 4hours
  Varies between 0-10 point (no pain- more severe pain) for patient self-reporting of pain for actual pain

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Kumru, MD PhD, Principal Investigator — Neurologist
Locations (1):
- Institut Guttmann, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No